CLINICAL TRIAL: NCT00916669
Title: A Randomized Phase II Study to Evaluate the Effect of Two Different Doses of Enoxaparin Sodium in Combination With Standard Chemotherapy (Cisplatin Plus Etoposide) With Respect to Time to Tumor Progression (TTP) in Patients With Newly Diagnosed Extensive Stage Small Cell Lung Cancer (SCLC) Without Underlying Venous Thromboembolism
Brief Title: A Randomized Study to Evaluate the Effect of Two Different Doses of Enoxaparin Sodium in Combination With Standard Chemotherapy in Patients With Stage Small Cell Lung Cancer (SCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor withdrew funding prior to patient enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); North Shore Medical Center (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Rachel P. Rosovsky, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-097
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2010-07

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; enoxaparin sodium; cisplatin; etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Cisplatin; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Active Comparator): Cisplatin and Etoposide
  Interventions: Drug: Etoposide; Drug: Cisplatin
- Group B (Experimental): Cisplatin and etoposide, plus low-dose enoxaparin sodium
  Interventions: Drug: Etoposide; Drug: Cisplatin; Drug: enoxaparin sodium
- Group C (Experimental): Cisplatin and etoposide, plus high-dose enoxaparin sodium
  Interventions: Drug: Etoposide; Drug: Cisplatin; Drug: enoxaparin sodium

INTERVENTIONS:
Drug: Etoposide — Etoposide given as an infusion on day 1, day 2 and day 3 of a three-week cycle for a total of 6 cycles
Drug: Cisplatin — Given as an infusion on day 1 of a three-week cycle for a total of 6 cycles
Drug: enoxaparin sodium — Given as a subcutaneous injection in the abdomen daily during chemotherapy treatment and then continuing daily for 1 year. Dose will vary.
  Other Names: Lovenox
  Arms: Group B; Group C

SUMMARY:
The purpose of this research study is to see if adding enoxaparin sodium to standard treatment with the chemotherapy drugs cisplatin and etoposide will help treat extensive stage SCLC. Two different doses of enoxaparin sodium will be studied in order to determine if one dose is more effective than the other. Enoxaparin sodium (Lovenox) is a drug that is approved by the FDA to help treat or prevent blood clots. Results from previous research studies suggest that adding enoxaparin sodium to standard treatment improved the response to treatment for some study participants with various types of cancer.

DETAILED DESCRIPTION:
* Since no one knows which of the study options are best, participants will be randomized into one of three study treatment groups. Group A will receive cisplatin and etoposide. Group B will receive cisplatin and etoposide plus low-dose enoxaparin sodium. Group C will receive cisplatin and etoposide plus high-dose enoxaparin sodium.
* Study treatment will be divided into chemotherapy and post-chemotherapy periods. All three groups (Group A, B and C) will receive six 3-week cycles of chemotherapy. Groups B and C will also receive daily enoxaparin sodium during the chemotherapy stage and daily enoxaparin sodium for 1 year after the chemotherapy.
* Cisplatin and etoposide are given as an infusion in 3-week cycles for up to six cycles. Enoxaparin sodium is given as an injection under the skin into the sides of the abdomen. Participants will be instructed in how to give themselves the injections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically or cytologically documented extensive disease small cell lung cancer. Only small cell histology is eligible. Mixed histology is not eligible. Patients who are considered to have operable disease are not eligible
* Radiographic measurable disease by RECIST criteria
* Life expectancy of greater than 4 months and ECOG Performance Status of less than or equal to 2
* Patients must be an appropriate candidate for the standard combination of cisplatin and etoposide for SCLC. There are no restrictions on radiotherapy
* No prior chemotherapy for SCLC cancer
* Participants must meet the hematological, renal and hepatic function requirements outlined in the protocol
* If brain or bone metastases are present at the time of initial diagnosis, patients must have completed radiation treatment at least 2 weeks before starting the study
* No active uncontrolled infection
* No other serious illness or medical condition that in the opinion of the investigator would be expected to interfere with the subject's ability to receive study treatment or comply with study procedures

Exclusion Criteria:

* New (defined as 6 months or less) or symptomatic thrombosis at the time of enrollment
* Indication for anticoagulant treatment such as mechanical heart valves, atrial fibrillation, or previous VTE
* Contraindication or known hypersensitivity to LMWH or unfractionated heparin (UFH)
* Active bleeding disorder
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding women
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers will are eligible if diagnosed and treated within the past 5 years; cervical in situ, and basal cell or squamous cell carcinoma of the skin
* HIV-positive individuals on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the prophylactic and treatment doses of Enoxaparin sodium given in combination with standard chemotherapy compared to standard chemotherapy alone with respect to time to tumor progression in this patient population. | 2 years

SECONDARY OUTCOMES:
To determine the effect of 2 different doses of enoxaparin sodium in combination with chemotherapy and chemotherapy alone on biomarkers of angiogenesis and to identify if these markers correlate with overall survival and progression free survival. | 2 years
To evaluate toxicity and determine the rates of bleeding complications in this patient population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rosovsky, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - North Shore Medical Center, Peabody, Massachusetts